CLINICAL TRIAL: NCT02725125
Title: Single-arm,Two Phase,Multicenter Trial to Evaluating the Efficacy and Safety of the CAR-T for Stomach Cancer
Brief Title: Study Evaluating the Efficacy and Safety With CAR-T for Stomach Cancer
Acronym: EECSC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sinobioway Cell Therapy Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACCO-2015-06-04
Record Dates: First submitted 2016-03-25; First posted 2016-03-31 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Stomach Neoplasms
Keywords: Stomach Cancer CAR-T
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single-arm (Experimental): Name:The Chimeric Antigen Receptor T Cell Immunotherapy (CAR-T) Dosage form：injection Dosage:100ml/time Frequency:0days,the first day,the second day,28 days,29 days Duration:total five times
  Interventions: Biological: EPCAM-targeted CAR-T cells

INTERVENTIONS:
Biological: EPCAM-targeted CAR-T cells — This study have only one arm that is CAR-T experimental arm. Firstly all participators will be attended the screening, who passed the screening for the treatment of CAR-T cells, the CAR-EPCAM-modified T cells can recognize and kill tumor cells in the body，follow-up 35 months.

SUMMARY:
This single-arm, multicenter Phase 2 trial will treat the patients who have relapsed or refractory stomach cancer with an infusion of the patient's own T cells that have been genetically modified to express a chimeric antigen receptor(CAR) that will bind to tumor cells that express the EPCAM protein on the cell surface.The study will determine if these modified T cells help the body's immune system eliminate tumor cells.The trial will also study the safety of treatment with CAR-T, how long CAR-T cells stay in the patient's body and the impact of this treatment on survival.

DETAILED DESCRIPTION:
This is a single-arm, multicenter Phase 2 study to evaluate the efficacy and safety of the CAR-T for Stomach Cancer. The study will be conducted using a phaseⅠ /Ⅱ design.The study will have the following sequential phases: Part A(screening leukapheresis, cell product preparation, and cytoreductive chemotherapy) and Part B(treatment and follow-up). The follow-up period for each participant is approximately 35 months after the final CAR-T infusion.The total duration of the study is expected to be approximately 3 years. A total of 19 patients may be enrolled over a period of 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. According to UICC or gastric cancer diagnosis and treatment guideline of diagnosis for patients with gastric cancer, first-line and second-line chemotherapy of advanced gastric cancer, and through flow cytometry or immune tissues (cell) chemistry, confirm the tumor cells positive expression of relevant molecular targets;
2. Age <=75 years old, both male and female;
3. Is expected to survive more than 3 months;
4. Physical condition is good: 0-2 score ECOG score;
5. The lymphocyte count must > =0.4*10^9/L at the time of collection of peripheral blood;
6. Vital organs (heart, kidney) function is normal, there is no major wound healing. No serious virus, bacterial infection;
7. Non pregnancy and lactation;
8. History of severe allergic reactions without biological products;
9. Voluntary participation, good compliance,the subjects can cooperate with the experimental observation, and signed a written Informed Consent Form;
10. At least one measurable lesion.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Organ failure, such as heart: Class III and IV; liver: to Chlid grading of liver function grade C; kidney: kidney failure and uremia stage; lung: symptoms of severe respiratory failure; brain: disorder of consciousness;
3. Patients with significant graft versus host disease (GVHD) after organ transplant history or allogeneic hematopoietic stem cell transplantation;
4. Long term use of immunosuppressive drugs or people with severe autoimmune diseases;
5. Any other chronic disease patients who have been treated with immune agents or hormone therapy;
6. A serious infectious disease with severe, uncontrollable, wound healing
7. Allergy to the interleukin and interferon cytokine;
8. Coagulation abnormalities and severe thrombosis;
9. Patients who have participated in other clinical trials or other clinical trials in the past 30 days
10. The Investigator believe the patients should not participate in this experiment.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2015-11; Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Disease control rates | 0 to 180 days

SECONDARY OUTCOMES:
Duration of remission | 0 to 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Yifu He, PI, Principal Investigator — Associate chief physician
Locations (1):
- Anhui Provincial Cancer Hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No
No plans to share data.